CLINICAL TRIAL: NCT03733132
Title: Metformin Effect on Brain Function in Insulin Resistant Elderly People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Professor of Medicine and Consultant in Endocrinology and Metabolism, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18-004012; 1R21AG060139-01 (NIH)
Record Dates: First submitted 2018-10-16; First posted 2018-11-07 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Insulin Resistance; Obesity; Obesity, Abdominal
Keywords: Insulin Resistance; Cognition; Cognitive Impairment; Brain Function
MeSH Terms: conditions — Insulin Resistance; Obesity; Obesity, Abdominal; Cognitive Dysfunction | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study will be a double-blind, placebo-controlled, randomized design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants in placebo group will receive Placebo Oral Tablets identical to the metformin tablets for 10 months.
  Interventions: Drug: Placebo Oral Tablet
- Metformin (Active Comparator): Participants in placebo group will receive an escalating dose of Metformin hydrochloride tablets up to a dose of 2500mg for 10 months.
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin treatment of 2500mg for 10 months in the Metformin group
  Other Names: Metformin
  Arms: Metformin
Drug: Placebo Oral Tablet — Placebo treatment of identical tablets to metformin group
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) and other forms of dementia are rapidly increasing with the aging of the population, and show a clear preponderance among people with insulin resistance. Metformin, an insulin sensitizer, is being examined in clinical trials as an anti-aging drug. However, very little objective data is available regarding metformin's effect on the brain, a major organ affected by aging.

DETAILED DESCRIPTION:
Insulin resistance is highly prevalent with advancing age. Metformin is an insulin sensitizer and is currently being extensively investigated for its potential anti-aging effect. However, only very limited information is available on metformin effect on brain, which is a major organ affected by aging. With appropriate experimental design, the investigators are attempting to understand the mechanism of metformin treatment on the physiology of the brain as well as cognitive effects. These studies may uncover relationships that could be favorably manipulated to decrease health risks associated with insulin sensitivity and the effect on the brain.

The study results may lead to a breakthrough in providing either definitive data or sufficiently strong preliminary data regarding metformin's effect on elderly people with insulin resistance, on whether the drug enhances brain mitochondrial function in conjunction with improvement of brain functional network and cognitive function.

The overall hypothesis is that metformin administration to elderly people with insulin resistance enhances brain mitochondrial function in conjunction with improvement of brain function. To test this hypothesis, the investigators will address the following Specific Aims:

1. Determine whether 40 weeks of metformin administration in elderly people (> 65 years) with insulin resistance enhances brain mitochondrial ATP production. The investigators will measure brain ATP production by 31P-MRS.
2. Determine the effect of 40 weeks of metformin administration in elderly people (> 65 years) with insulin resistance on blood flow and functional network in different areas of brain. As a secondary outcome, the investigators will measure structural changes in white and grey matter areas of brain to determine whether metformin has any effect on brain structure.
3. Determine the effect of 40 weeks of metformin administration in elderly people (> 65 years) with insulin resistance on cognitive function. The investigators will utilize the computerized NIH Toolbox to measure cognitive outcomes.

The investigators will also associate outcomes from our specific aims with improvements in whole-body insulin sensitivity and skeletal muscle mitochondrial function.

The investigators propose to complete 40 weeks of study in 40 elderly (> 65 years) participants with fasting glucose between 100 to 140 mg/dl and abdominal girth of >102 cm in men and > 88 cm in women. All participants will be those who are not oral hypoglycemic agents including metformin. In this double-blind placebo trial, the investigators will randomly assign the participants to placebo or metformin in an escalated dose to reach a maximum of 2500 mg per day.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 65 years
* Abdominal girth > 102 cm in men and > 88 cm in women-
* Fasting glucose >/= 100-140 mg/dL
* Non-smoker
* English language proficiency

Exclusion Criteria:

* Coronary artery disease or heart failure
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

Inpatient psychiatric treatment in the past 6 months

* Presence of a known adrenal disorder
* Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
* Abnormal renal function tests results (calculated GFR <60 mL/min/1.73m2); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty
* Active gastroparesis
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
* Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L): testing required within here months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise
* Abuse of alcohol or recreational drugs
* Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis)
* Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg) at the time of screening
* Oral steroids
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
* Any metal in the body that could interfere with magnetic resonance imaging (MRI) including pacemaker or implanted defibrillator, neurostimulators, ear implants, metal fragments within the body, metal joints, rods, pins, plates or screws
* Medications that may impact study end points such as mitochondrial biology eg. beta blockers
* Anti-hyperglycemic drugs including metformin
* Any other medication that the investigator believes is a contraindication to the subject's participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Sreekumaran Nair, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants in the placebo group received Placebo Oral Tablets identical to the metformin tablets for 10 months.
  Placebo Oral Tablet: Placebo treatment of identical tablets to metformin group
- Metformin: Participants in Metformin group received an escalating dose of Metformin hydrochloride tablets up to a dose of 2500mg for 10 months.
  Metformin Hydrochloride: Metformin treatment of 2500mg for 10 months in the Metformin group
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.006 (4.083) | 67.584 (5.375) | 67.295 (4.720)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 12 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 20 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brain PCr/ATP Ratio as Measured by Phosphorus Magnetic Spectroscopy (31P-MRS) After 10 Months of Metformin Administration
Description: Multivoxel spectroscopic imaging of the brain will be performed using our dual-tuned single-channel-proton eight-channel-phosphorus head coil. A single 2.5 cm thick slice will be prescribed to encompass the temporal and occipital lobes, and weighted MRSI will be performed using a 16x16 matrix to acquire nominal 2.5 cm3 voxels. Multivoxel phosphorus magnetic resonance spectroscopic imaging data were reconstructed and quantified using jMRUI 6.0. Spectra were preprocessed by (a) truncating the data to 768 points, then 0-filling to 1024 points; (b) apodizing with a 5 Hz Lorenzian; and (c) aligning the data such that the PCr peak was set to 0 Hz. Next, 2 voxels from occipital lobe were selected, extracted, and averaged together into a single free induction decay in order to reduce noise. The outcome measure PCr/ATP ratio is a marker of ATP resynthesis potential and is reported as a change from pre- to post-treatment.
Time Frame: Baseline, 10 months
Population: If PCr, γ-ATP, α-ATP, or β-ATP signals were indiscernible from the background noise after processing then those spectra were discarded. Spectra processing was performed by one person, and processing steps were checked for fidelity by a second person. Twelve patients in the placebo group and 15 in the metformin group meet quality control criteria for both the pre- and post-scans.
Measure: Mean (Standard Deviation); unit: PCr/ATP ratio
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 12 | 15
PCr/ATP ratio | -0.045 (0.258) | -0.016 (0.483)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority; p = 0.854, t-test, 2 sided

2. Primary Outcome: Change From Baseline in Cognitive Function as Measured by NIH Toolbox After 10 Months of Metformin Administration
Description: The NIH Toolbox will be utilized to measure cognitive outcomes. The NIH Toolbox-Cognition Battery is composed of 7 tests (~30 minutes) and our primary outcome measure will be the Total Cognition Composite score comprised from these 7 tests. Results are presented as a fully-adjusted T-score. For a single timepoint, T-scores are expected to have a population mean of 50, standard deviation of 10. For a single timepoint, higher T-scores indicate better cognitive test performance. An increase in T-score over time is considered a better outcome. At the individual level, a T-score < 40 is considered low test performance. There were no clear clinically relevant thresholds for a change in T-score over 10 months at the start of this study. Comparison of the mean change in T-score over time in the Metformin treatment group to placebo is our analysis of interest
Time Frame: Baseline, 10 months
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 20 | 20
t-score | 1.450 (4.968) | 2.900 (5.543)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority; p = 0.389, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Brain Structure as Measured by MRI After 10 Months of Metformin Administration
Description: AA sagittal 3D MPRAGE sequence with 0.7mm isotropic voxels (TR=2400, TE=2.57, TI=1100, FA=8) will be used to acquire high-resolution structural data for volumetric analysis of brain region changes related to metformin. To measure white matter information: An axial 2D symmetric multi-slice (SMS) diffusion tensor imaging (DTI) sequence with 60 diffusion directions, 5 B0 acquisitions and 2mm isotropic voxels (TR=3000, TE=73, FA=90, ETL 43, both A-P and P-A phase encoding for B0 images) will be used to acquire white matter integrity data related to metformin.
Time Frame: Baseline, 10 months
Population: One participant in each group was not able to be analyzed due to lack of sufficent scan quality.
Measure: Mean (Standard Deviation); unit: mm cubed
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 19 | 19
mm cubed | -2255.098 (11757.866) | 1588.247 (30282.932)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority; p = 0.609, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Muscle Mitochondrial Respiration as Measured by High-resolution Respirometry Following 10 Months of Metformin Administration
Description: High-resolution respirometry will be used to analyze oxygen consumption in isolated mitochondria from skeletal muscle biopsy samples while simultaneously quantifying reactive oxygen species (ROS) production using amplex red. An increase in mitochondrial respiration is indicative of increased mitochondrial function which is a positive outcome.
Time Frame: Baseline, 10 months
Population: 2 participants in each group were unable to be measured for mitochondrial respiration. 2 were due to instrumentation malfunction and 2 were due to inability to collect enough muscle tissue for mitochondrial isolation on one or both study dates.
Measure: Mean (Standard Deviation); unit: pmol/sec/mL/mg tissue mass
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 18 | 18
pmol/sec/mL/mg tissue mass | -0.106 (2.752) | -0.926 (2.674)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority; p = 0.371, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Muscle Mitochondrial ATP Production as Measured by Fluorometry Following 10 Months of Metformin Administration
Description: Concurrent to mitochondrial respiration, muscle mitochondrial ATP production will be measured using high-sensitivity fluorometry. An increase in mitochondrial ATP production shows increase mitochondrial efficiency which is a positive outcome.
Time Frame: Baseline, 10 months
Population: 5 participants in the placebo group and 6 in the metfomin group were unable to be analyzed. One in each group was due to the inability to collect enough muscle for mitochondrial isolation and the remainder were due to an equipment breakdown (power source - had to be externally source and repaired via service technician) that rendered the equipment unusable for multiple study days.
Measure: Mean (Standard Deviation); unit: pmol/sec/ug mitochondrial protein
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 15 | 14
pmol/sec/ug mitochondrial protein | 5.760 (13.218) | 8.899 (26.430)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority; p = 0.686, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Placebo | Metformin
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Metformin (N=20)
COVID-19 infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Metformin (N=20)
Infections and infestations: Other (Infections and infestations) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 7 (8)
Social circumstances (Social circumstances) | 0 (0) | 1 (1)
Eye disorders (Eye disorders) | 1 (1) | 0 (0)
COVID-19 Infection (Infections and infestations) | 2 (2) | 1 (1)
Nausea (General disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Weight loss (General disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03733132/Prot_SAP_ICF_001.pdf